CLINICAL TRIAL: NCT02539225
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Study of S-1 and Oxaliplatin With or Without Ramucirumab as First-line Therapy Followed by Paclitaxel With Ramucirumab as Second-line Therapy in Patients With Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: A Study of Ramucirumab in Participants With Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15461; I4T-JE-JVCW (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Metastatic Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Ramucirumab; S 1 (combination); Oxaliplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-1/Oxaliplatin + Ramucirumab (Experimental): (Part A) Ramucirumab intravenously (IV) on day 1 and day 8 along with S-1 by mouth (PO) on days 1-14 and oxaliplatin IV on day 1 of each 21 day cycle. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criterion is met then move to Part B.
  (Part B) Ramucirumab IV on day 1 and day 15 along with paclitaxel IV on day 1, 8, and 15 of each 28 day cycle. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criterion is met.
  Interventions: Drug: Ramucirumab; Drug: S-1; Drug: Oxaliplatin; Drug: Paclitaxel
- S-1/Oxaliplatin + Placebo (Active Comparator): (Part A) Placebo IV on day 1 and day 8 along with S-1 PO on days 1-14 and oxaliplatin IV on day 1 of each 21 day cycle. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criterion is met then move to Part B.
  (Part B) Ramucirumab IV on day 1 and day 15 along with paclitaxel IV on day 1, 8, and 15 of each 28 day cycle. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criterion is met.
  Interventions: Drug: Ramucirumab; Drug: Placebo; Drug: S-1; Drug: Oxaliplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806; IMC-1121B; Cyramza
Drug: Placebo — Administered IV
  Arms: S-1/Oxaliplatin + Placebo
Drug: S-1 — Administered PO
Drug: Oxaliplatin — Administered IV
Drug: Paclitaxel — Administered IV

SUMMARY:
The main purpose of this study is to evaluate the effectiveness of S-1 and oxaliplatin with or without ramucirumab as first line therapy in participants with metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Have a histopathologically or cytologically confirmed diagnosis of metastatic gastric or GEJ adenocarcinoma. Participants with esophageal cancer are not eligible.
* Have not received any prior first-line systemic therapy for gastric or GEJ adenocarcinoma (prior adjuvant or neoadjuvant therapy is permitted). Participants whose disease has progressed after >24 weeks following the last dose of systemic treatment in the adjuvant/neoadjuvant setting are eligible.
* Have measurable or nonmeasurable but evaluable disease determined using guidelines in Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v.1.1).
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale at baseline.
* Have adequate organ function.
* Have an estimated life expectancy of ≥12 weeks in the judgment of the investigator.
* Eligible participants of reproductive potential (both sexes) must agree to use contraception (hormonal or barrier methods) during the study period and at least 6 months after the last dose of study treatment or longer if required per local regulations.
* Are willing to provide a blood sample for research purposes. Submission of a blood sample is mandatory for participation in this study unless restricted by local regulations or ethical review boards (ERBs); submission of a tumor tissue sample is optional.

Exclusion Criteria:

* Participants with human epidermal growth factor receptor 2 (HER2)-positive status as determined per local standards. Participants with a negative test or having an indeterminate result due to any reason are eligible, provided these participants are not eligible for treatment directed against tumors which overexpress HER2.
* Have radiation therapy within 14 days prior to randomization. Any lesion requiring palliative radiation or which has been previously irradiated cannot be considered for response assessment.
* Have documented brain metastases, leptomeningeal disease, or uncontrolled spinal cord compression.
* Have undergone major surgery within 28 days prior to randomization.
* Are currently enrolled in, or discontinued study drug within the last 28 days from, a clinical trial involving an investigational product or non-approved use of a drug or device (other than the study drug used in this study), or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study. Participants participating in surveys or observational studies are eligible to participate in this study.
* Are pregnant or breast feeding. Females of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to first dose of study treatment.
* Have any prior malignancies.
* Have any condition (eg, psychological, geographical, or medical) that does not permit compliance with the study and follow-up procedures or suggest that the participant is, in the investigator's opinion, not an appropriate candidate for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (24):
- Japan (18):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Akashi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bunkyō City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gifu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kōtoku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagoya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sagamihara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sakai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sapporo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shinjuku-Ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suita-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Takatsuki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Toyonaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Utsunomiya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yokohama
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulsan
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuei Shan Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Yoshikawa T, Muro K, Shitara K, Oh DY, Kang YK, Chung HC, Kudo T, Chin K, Kadowaki S, Hamamoto Y, Hironaka S, Yoshida K, Yen CJ, Omuro Y, Bai LY, Maeda K, Ozeki A, Yoshikawa R, Kitagawa Y. Effect of First-line S-1 Plus Oxaliplatin With or Without Ramucirumab Followed by Paclitaxel Plus Ramucirumab on Advanced Gastric Cancer in East Asia: The Phase 2 RAINSTORM Randomized Clinical Trial. JAMA Netw Open. 2019 Aug 2;2(8):e198243. doi: 10.1001/jamanetworkopen.2019.8243. PMID 31373648
- See also: A Study of Ramucirumab in Participants With Gastric or Gastroesophageal Junction Adenocarcinoma — https://trials.lillytrialguide.com/en-US/trial/1iuJn3anbEq6WK6y64aEY4

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Completers are defined as participants who died or those who were alive and off treatment at study completion.
Groups:
- Ramucirumab + S-1 + Oxaliplatin: Part A: Participants received 8 milligram per kilogram (mg/kg) Ramucirumab by intravenous (IV) infusion on day 1 and day 8 of 21 days cycle in combination with oral dose of 80-120 mg/day S-1 on days 1 to14 and 100 milligram per square meter (mg/m^2) Oxaliplatin administered by IV infusion on day 1 until disease progression or any other discontinuation criteria is met.
  Part B:Participants received 8 mg/kg Ramucirumab by intravenous infusion on day 1 and day 15 of 28 days cycle in combination with 80 mg/m^2 Paclitaxel on day 1, 8 and 15 by intravenous infusion until disease progression or any other discontinuation criteria is met.
- Placebo + S-1 + Oxaliplatin: Part A: Participants received placebo by intravenous (IV) infusion on day 1 and day 8 of 21 days cycle in combination with oral dose of 80-120 mg/day S-1 on days 1 to14 and 100 milligram per square meter (mg/m^2) Oxaliplatin administered by IV infusion on day 1 until disease progression or any other discontinuation criteria is met.
  Part B:Participants received Ramucirumab by intravenous infusion on day 1 and day 15 of 28 days cycle in combination with 80 mg/m^2 Paclitaxel on day 1, 8 and 15 by intravenous infusion until disease progression or any other discontinuation criteria is met.
Period: Part A
Arm/Group | Ramucirumab + S-1 + Oxaliplatin | Placebo + S-1 + Oxaliplatin
Started | 97 | 94
Received Any Quantity of Study Drug | 96 | 93
Completed | 77 | 78
Not Completed | 20 | 16
Not completed — Adverse Event | 13 | 4
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Physician Decision | 4 | 7
Not completed — Did Not Receive study Drug | 1 | 1
Period: Pre Treatment for Part B
Arm/Group | Ramucirumab + S-1 + Oxaliplatin | Placebo + S-1 + Oxaliplatin
Started | 63 (Participants who met initiation criteria of Part B were allowed to pretreatment for part B.) | 66 (Participants who met initiation criteria of Part B were allowed to pretreatment for part B.)
Completed | 58 | 64
Not Completed | 5 | 2
Not completed — Progressive disease | 1 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 2 | 0
Period: Part B
Arm/Group | Ramucirumab + S-1 + Oxaliplatin | Placebo + S-1 + Oxaliplatin
Started | 58 | 64
Completed | 54 | 48
Not Completed | 4 | 16
Not completed — Adverse Event | 4 | 4
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Physician Decision | 0 | 9

BASELINE CHARACTERISTICS:
Population: All randomized participants who received any quantity of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramucirumab + S-1 + Oxaliplatin | Placebo + S-1 + Oxaliplatin | Total
Number analyzed (Participants) | 96 | 93 | 189
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.2 (12.35) | 61.3 (11.53) | 60.2 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 29 | 68
  Male | 57 | 64 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 96 | 93 | 189
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 96 | 93 | 189
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 20 | 20 | 40
  Japan | 65 | 64 | 129
  Taiwan | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization until the date of objectively determined progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) or death from any cause, whichever is first. Disease progression is defined as ≥20% increase in the sum of diameters of target lesions, taking as reference smallest sum on study (included baseline sum if that was the smallest on study); sum must have demonstrated an absolute increase of ≥5 millimeter (mm) or the appearance of ≥1 new lesions was progression. Participants who did not progress, were lost to follow-up were censored at the day of their last adequate tumor assessment.
Time Frame: Randomization to Radiographic Documentation of Progression or Death Due to Any Cause (Up to 25 Months)
Population: All randomized participants who received any quantity of study drug in Part A. Censored participants: Ramucirumab + S-1 + Oxaliplatin = 23; Placebo + S-1 + Oxaliplatin = 19.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Ramucirumab + S-1 + Oxaliplatin | Placebo + S-1 + Oxaliplatin
Number analyzed (Participants) | 96 | 93
Months | 6.34 [5.65 to 6.93] | 6.74 [5.75 to 7.13]
Statistical Analysis 1: Comparison: Ramucirumab + S-1 + Oxaliplatin vs Placebo + S-1 + Oxaliplatin; Test type: Superiority; p = 0.698, Stratified Log Rank

2. Secondary Outcome: Progression-free Survival to the Second Disease Progression (PFS 2)
Description: Progression-free survival 2 (PFS2) is defined as the time from the date of randomization to second disease progression (defined as the date of first tumor assessment observing PD defined by RECIST v.1.1, after the start of second-line therapy using the last tumor assessment before starting the second-line therapy (RAM+PTX) as the baseline assessment), or death of any cause, whichever occurs first. If the second-line therapy was not started, the OS will be substituted for PFS2. If a post-discontinuation therapy was started before observing PD after the start of second-line therapy. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. PFS2 will be censored at the date of the last adequate tumor assessment on or before staring the post-discontinuation therapy.
Time Frame: Randomization to Second Radiographic Documentation of Progression or Death Due to Any Cause (Up to 31 Months)
Population: All randomized participants who received any quantity of study drug. Censored participants: Ramucirumab + S-1 + Oxaliplatin = 26; Placebo + S-1 + Oxaliplatin = 26.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Ramucirumab + S-1 + Oxaliplatin | Placebo + S-1 + Oxaliplatin
Number analyzed (Participants) | 96 | 93
Months | 10.94 [9.63 to 12.52] | 11.99 [9.82 to 13.83]
Statistical Analysis 1: Comparison: Ramucirumab + S-1 + Oxaliplatin vs Placebo + S-1 + Oxaliplatin; Test type: Superiority; p = 0.549, Log Rank Stratified

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as time from the date of randomization to the date of death from any cause. If the patient was alive at the cut-off for analysis (or lost to follow-up), OS data were censored for analysis on the last date the patient was known to be alive.
Time Frame: Randomization to Death Due to Any Cause (Up to 31 Months)
Population: All randomized participants who received at least one dose of study drug. Censored participants: Ramucirumab + S-1 + Oxaliplatin = 27; Placebo + S-1 + Oxaliplatin = 30.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Ramucirumab + S-1 + Oxaliplatin | Placebo + S-1 + Oxaliplatin
Number analyzed (Participants) | 96 | 93
Months | 14.65 [12.39 to 15.67] | 14.26 [13.83 to 17.31]
Statistical Analysis 1: Comparison: Ramucirumab + S-1 + Oxaliplatin vs Placebo + S-1 + Oxaliplatin; Test type: Superiority; p = 0.548, Log Rank Stratified

4. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR)
Description: The ORR is the number of all participants with Partial Response (PR) or Complete Response (CR) according to RECIST v1.1 from the start of the treatment until disease progression/recurrence. CR is defined as the disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 mm. PR is defined as ≥30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph nodes), taking as reference the baseline sum diameter. Disease progression is defined as ≥20% increase in the sum of diameters of target lesions, taking as reference smallest sum on study (included baseline sum if that was the smallest on study); sum must have demonstrated an absolute increase of ≥5 mm or the appearance of ≥1 new lesions was progression.
Time Frame: Randomization to Disease Progression (Up to 25 Months)
Population: All randomized participants who received any quantity of study drug in Part A with measurable disease.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab + S-1 + Oxaliplatin | Placebo + S-1 + Oxaliplatin
Number analyzed (Participants) | 55 | 54
percentage of participants | 58.2 [49.7 to 66.7] | 50.0 [41.3 to 58.7]
Statistical Analysis 1: Comparison: Ramucirumab + S-1 + Oxaliplatin vs Placebo + S-1 + Oxaliplatin; Test type: Superiority; p = 0.402, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.374, 80% CI 2-sided [0.844 to 2.236]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) was the percentage of participants with a best overall response of CR, PR, or Stable Disease (SD) as per Response using RECIST v1.1 criteria. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions. Disease progression is defined as ≥20% increase in the sum of diameters of target lesions, taking as reference smallest sum on study (included baseline sum if that was the smallest on study); sum must have demonstrated an absolute increase of ≥5 mm or the appearance of ≥1 new lesions was progression.
Time Frame: Randomization to Disease Progression (Up to 25 Months)
Population: All randomized participants who received any quantity of study drug in Part A with measurable disease.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab + S-1 + Oxaliplatin | Placebo + S-1 + Oxaliplatin
Number analyzed (Participants) | 55 | 54
percentage of participants | 90.9 [85.9 to 95.9] | 87 [81.2 to 92.9]
Statistical Analysis 1: Comparison: Ramucirumab + S-1 + Oxaliplatin vs Placebo + S-1 + Oxaliplatin; Test type: Superiority; p = 0.501, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.527, 80% CI 2-sided [0.680 to 3.433]

6. Secondary Outcome: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Ramucirumab in Part A
Description: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Ramucirumab in Part A.
Time Frame: Cycle 1 Day 1 & 8 Predose, Cycle 2 Day 1 Predose, Cycle 3 Day 1 Predose, Cycle 5 Day 1 Predose, Cycle 9 Day 1 Predose
Population: All randomized participants who received at least one dose of ramucirumab in part A and had evaluable PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (ug/mL)
Groups:
- Ramucirumab + S-1 + Oxaliplatin - Part A: Participants received 8 milligram per kilogram (mg/kg) Ramucirumab by intravenous (IV) infusion on day 1 and day 8 of 21 days cycle in combination with oral dose of 80-120 mg/day S-1 on days 1 to14 and 100 milligram per square meter (mg/m^2) Oxaliplatin administered by IV infusion on day 1 until disease progression or any other discontinuation criteria is met.
Arm/Group | Ramucirumab + S-1 + Oxaliplatin - Part A
Number analyzed (Participants) | 96
Microgram per milliliter (ug/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 94
  Cycle 1 Day 1 | NA (NA) — Samples for Ramucirumab group at cycle 1 day 1 were below the limit of quantification and treated as missing for analysis.
  Cycle 1 Day 8: number analyzed (Participants) | 91
  Cycle 1 Day 8 | 42.6 (32)
  Cycle 2 Day 1: number analyzed (Participants) | 85
  Cycle 2 Day 1 | 41.4 (40)
  Cycle 3 Day 1: number analyzed (Participants) | 68
  Cycle 3 Day 1 | 59.4 (51)
  Cycle 5 Day 1: number analyzed (Participants) | 38
  Cycle 5 Day 1 | 83.6 (37)
  Cycle 9 Day 1: number analyzed (Participants) | 15
  Cycle 9 Day 1 | 94.6 (38)

7. Secondary Outcome: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Ramucirumab in Part B
Description: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Ramucirumab in Part B.
Time Frame: Cycle 1 Day 1 predose, Cycle 2 Day 1 predose
Population: All randomized participants who received at least one dose of ramucirumab in part B and had evaluable PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (ug/mL)
Groups:
- Ramucirumab + S-1 + Oxaliplatin Part B: Participants received 8 mg/kg Ramucirumab by intravenous infusion on day 1 and day 15 of 28 days cycle in combination with 80 mg/m^2 Paclitaxel on day 1, 8 and 15 by intravenous infusion until disease progression or any other discontinuation criteria is met.
- Placebo + S-1 + Oxaliplatin - Part B: Participants received Ramucirumab by intravenous infusion on day 1 and day 15 of 28 days cycle in combination with 80 mg/m^2 Paclitaxel on day 1, 8 and 15 by intravenous infusion until disease progression or any other discontinuation criteria is met.
Arm/Group | Ramucirumab + S-1 + Oxaliplatin Part B | Placebo + S-1 + Oxaliplatin - Part B
Number analyzed (Participants) | 58 | 64
Microgram per milliliter (ug/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 43 | 53
  Cycle 1 Day 1 | 52.0 (65) | NA (NA) — Samples for placebo group were below the limit of quantification and treated as missing for analysis
  Cycle 2 Day 1: number analyzed (Participants) | 29 | 38
  Cycle 2 Day 1 | 58.1 (40) | 41.0 (45)

8. Secondary Outcome: Number of Participants With Anti-Ramucirumab Antibodies
Description: Participant is considered as treatment emergent anti-drug antibody (TE ADA) positive if the participant has at least one post baseline titer that is a 4-fold or greater increase in titer from baseline measurement. If baseline result is ADA Not Present, then the participant is TE ADA+ if there is at least one post baseline result of ADA Present with titer >= 20.
Time Frame: Baseline through 25 months
Population: All randomized participants who received any quantity of study drug in part A and had at least one baseline & post baseline antibody (ADA) measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + S-1 + Oxaliplatin | Placebo + S-1 + Oxaliplatin
Number analyzed (Participants) | 92 | 90
Participants | 1 | 3

ADVERSE EVENTS:
Time Frame: Up to 31 Months
Description: All randomized participants who received at least one dose of study drug. Adverse events data for pre-treatment Part B were included in part A.
  There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Groups:
- Placebo + S-1 + Oxaliplatin - Part A: Participants received placebo by intravenous (IV) infusion on day 1 and day 8 of 21 days cycle in combination with oral dose of 80-120 mg/day S-1 on days 1 to14 and 100 milligram per square meter (mg/m^2) Oxaliplatin administered by IV infusion on day 1 until disease progression or any other discontinuation criteria is met.
Arm/Group | Ramucirumab + S-1 + Oxaliplatin - Part A | Placebo + S-1 + Oxaliplatin - Part A | Ramucirumab + S-1 + Oxaliplatin Part B | Placebo + S-1 + Oxaliplatin - Part B
All-Cause Mortality (participants affected / at risk) | 2/96 | 1/93 | 1/58 | 0/64
Serious Adverse Events (participants affected / at risk) | 29/96 | 24/93 | 16/58 | 14/64
Other Adverse Events (participants affected / at risk) | 95/96 | 93/93 | 58/58 | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + S-1 + Oxaliplatin - Part A (N=96) | Placebo + S-1 + Oxaliplatin - Part A (N=93) | Ramucirumab + S-1 + Oxaliplatin Part B (N=58) | Placebo + S-1 + Oxaliplatin - Part B (N=64)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Gastric stenosis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Prepyloric stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystocholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mycobacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ramucirumab + S-1 + Oxaliplatin - Part A (N=96) | Placebo + S-1 + Oxaliplatin - Part A (N=93) | Ramucirumab + S-1 + Oxaliplatin Part B (N=58) | Placebo + S-1 + Oxaliplatin - Part B (N=64)
Anaemia (Blood and lymphatic system disorders) | 25 (37) | 20 (32) | 15 (19) | 11 (23)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (7) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 6 (17) | 6 (20) | 3 (9) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (13) | 2 (5) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (4) | 2 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1/34 (1) | 0 (0)
Eustachian tube patulous (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corneal erosion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hyalosis asteroid (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 5 (5) | 4 (4) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panophthalmitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Scleral haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 6 (6) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 11 (11) | 11 (12) | 2 (3) | 3 (6)
Abdominal pain (Gastrointestinal disorders) | 18 (26) | 21 (28) | 7 (7) | 4 (4)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 9 (11) | 6 (6) | 1 (1) | 5 (5)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 7 (7) | 6 (6) | 2 (2) | 5 (5)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 33 (52) | 30 (32) | 3 (3) | 6 (6)
Dental caries (Gastrointestinal disorders) | 2 (2) | 1 (2) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 49 (103) | 28 (62) | 10 (15) | 8 (10)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 4 (4) | 1 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 4 (4) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 4 (6) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 54 (90) | 37 (69) | 5 (5) | 4 (4)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary gland fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 27 (48) | 18 (25) | 9 (10) | 9 (9)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (5) | 3 (3) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 28 (49) | 21 (34) | 5 (6) | 7 (8)
Asthenia (General disorders) | 3 (4) | 2 (2) | 0 (0) | 5 (6)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
Face oedema (General disorders) | 3 (3) | 2 (2) | 3 (3) | 2 (2)
Fatigue (General disorders) | 28 (35) | 22 (35) | 7 (8) | 8 (9)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 2 (3) | 2 (4) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Infusion site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 6 (10) | 8 (17) | 1 (1) | 0 (0)
Injury associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 26 (35) | 20 (25) | 9 (11) | 7 (9)
Medical device site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nodule (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (4) | 0 (0) | 1 (1) | 1 (1)
Oedema (General disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (3)
Oedema peripheral (General disorders) | 26 (31) | 19 (24) | 8 (8) | 8 (8)
Pain (General disorders) | 8 (9) | 4 (4) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 22 (28) | 22 (43) | 7 (9) | 11 (15)
Sensation of foreign body (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenderness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (3) | 5 (5) | 2 (2) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Actinomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angular cheilitis (Infections and infestations) | 2 (2) | 2 (5) | 1 (3) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Cystitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 3 (5) | 0 (0) | 2 (2)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mycobacterial infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (4) | 4 (4) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Pharyngitis (Infections and infestations) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Purulence (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 8 (11) | 6 (7) | 3 (3) | 2 (2)
Urethritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 3 (6) | 2 (2) | 2 (2)
Wound infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 6 (13) | 1 (1) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (6) | 3 (4) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stoma site discharge (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 21 (32) | 12 (18) | 4 (6) | 3 (4)
Amylase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 25 (45) | 15 (26) | 5 (7) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 10 (11) | 7 (8) | 5 (8) | 4 (4)
Blood bilirubin increased (Investigations) | 2 (3) | 9 (11) | 3 (3) | 3 (5)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 3 (5) | 0 (0) | 2 (2) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endoscopic retrograde cholangiopancreatography (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 7 (9) | 5 (5) | 2 (2) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 3 (7) | 2 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 48 (156) | 32 (79) | 33 (85) | 36 (108)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritoneal effluent erythrocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 33 (67) | 28 (62) | 4 (4) | 4 (6)
Weight decreased (Investigations) | 11 (13) | 9 (18) | 3 (5) | 7 (8)
Weight increased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 24 (74) | 18 (58) | 19 (49) | 24 (59)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 53 (78) | 57 (90) | 9 (9) | 12 (12)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 2 (4) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (11) | 7 (12) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (11) | 3 (5) | 3 (3) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 1 (4) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 (14) | 11 (12) | 6 (10) | 10 (10)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (6) | 1 (1) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (8) | 2 (4) | 5 (6) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 6 (7) | 4 (4)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (13) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (9) | 3 (3) | 4 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 10 (11) | 3 (5) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (6) | 4 (4) | 7 (15)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (5) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/39 (1) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1/29 (1) | 0 (0) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 7 (7) | 5 (5) | 4 (4)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1/29 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 7 (8) | 6 (7) | 2 (2) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 21 (24) | 20 (20) | 5 (5) | 3 (3)
Headache (Nervous system disorders) | 16 (29) | 12 (21) | 1 (1) | 4 (5)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 5 (6) | 1 (1) | 0 (0) | 1 (2)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 7 (13) | 4 (4) | 3 (3) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 56 (88) | 70 (120) | 8 (8) | 14 (14)
Somnolence (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 10 (10) | 10 (11) | 6 (6) | 4 (4)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 5 (7) | 5 (5) | 0 (0) | 1 (2)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 25 (40) | 14 (25) | 6 (14) | 7 (10)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/57 (1) | 1/64 (1) | 0 (0) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penile oedema (Reproductive system and breast disorders) | 1/57 (1) | 0 (0) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1/57 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1/39 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1/29 (3) | 0 (0) | 0 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1/39 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 10 (12) | 3 (3) | 5 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 (34) | 6 (7) | 10 (10) | 14 (22)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 5 (6) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pleural adhesion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (12) | 2 (2) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (5) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10) | 2 (2) | 26 (26) | 30 (30)
Cutaneous symptom (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (10) | 5 (5) | 2 (2) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 15 (16) | 7 (7) | 2 (2) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (10) | 5 (7) | 3 (3) | 6 (6)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (10) | 1 (1) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 4 (4) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 17 (17) | 15 (15) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal cavity drainage (Surgical and medical procedures) | 2 (3) | 1 (1) | 2 (2) | 2 (3)
Bile duct stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cell-free and concentrated ascites reinfusion therapy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cerebrospinal fluid reservoir placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colostomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenterostomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal tube insertion (Surgical and medical procedures) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Haematoma evacuation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 0 (0) | 1/29 (1) | 0 (0) | 0 (0)
Ileostomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laparoscopic surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laparotomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrostomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal dilation procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Omental flap operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Omental implantation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 0 (0) | 1/29 (1) | 0 (0) | 0 (0)
Small intestinal intussusception reduction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stent placement (Surgical and medical procedures) | 2 (3) | 3 (3) | 1 (1) | 0 (0)
Suture insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thoracic cavity drainage (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureteral stent insertion (Surgical and medical procedures) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 28 (28) | 12 (13) | 1 (1) | 10 (11)
Hypotension (Vascular disorders) | 2 (2) | 4 (6) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular pain (Vascular disorders) | 3 (7) | 3 (3) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 2 (2) | 4 (8) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-08-29): https://cdn.clinicaltrials.gov/large-docs/25/NCT02539225/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT02539225/SAP_001.pdf